CLINICAL TRIAL: NCT00002140
Title: A Randomized, Double-Blind, Comparative Study of Azithromycin Versus Clarithromycin in Combination With Ethambutol for the Treatment of Disseminated Mycobacterium Avium Complex (MAC) Infection in AIDs Patients
Status: Completed | Phase: Phase 3 | Type: Interventional
Sponsor: Pfizer (Industry)
Organization: NIH AIDS Clinical Trials Information Service (Industry)
Masking: Double | Purpose: Treatment
Other Study IDs: 226B; 066-189; 189/189B
Record Dates: First submitted 1999-11-02; First posted 2001-08-31 (Estimated); Last update posted 2005-06-24 (Estimated); Status verified 1998-07

CONDITIONS: Mycobacterium Avium-intracellulare Infection; HIV Infections
Keywords: Mycobacterium avium-intracellulare Infection; Drug Therapy, Combination; Ethambutol; Acquired Immunodeficiency Syndrome; Azithromycin; Clarithromycin
MeSH Terms: conditions — Mycobacterium avium-intracellulare Infection; HIV Infections; Acquired Immunodeficiency Syndrome | interventions — Ethambutol; Clarithromycin; Azithromycin

INTERVENTIONS:
Drug: Ethambutol hydrochloride
Drug: Clarithromycin
Drug: Azithromycin

SUMMARY:
To evaluate the efficacy and safety of two different doses of azithromycin in combination with ethambutol for the treatment of patients with Mycobacterium avium complex (MAC) infection, and to determine whether an azithromycin-containing regimen is at least as safe and effective as the same regimen containing clarithromycin..

DETAILED DESCRIPTION:
Patients are randomized to receive azithromycin at one of two doses in combination with ethambutol or clarithromycin in combination with ethambutol for 24 weeks, after which they are evaluated for entry into a maintenance phase of treatment. Clinical, microbiologic, and safety assessments are performed every 3 weeks for the first 12 weeks, then monthly for the remaining 12 weeks.

ELIGIBILITY:
Inclusion Criteria

Patients must have:

* HIV seropositivity.
* Disseminated MAC.
* No MAC therapy between time of last positive blood culture draw and study entry (single-agent prophylaxis allowed).
* Life expectancy of at least 2 months.
* Consent of parent or guardian if below legal age of consent.

Exclusion Criteria

Co-existing Condition:

Patients with the following symptoms or conditions are excluded:

* Known hypersensitivity to macrolide antibiotics (erythromycin, azithromycin, or clarithromycin) or ethambutol.
* Inability to take oral medications.
* Condition likely to interfere with drug absorption (e.g., gastrectomy, malabsorption syndromes).

Concurrent Medication:

Excluded:

* Another investigational drug started in the week prior to study entry.

Prior Medication:

Excluded:

* MAC therapy between time of last positive blood culture draw and study entry (although single-agent prophylaxis is allowed).

Min Age: 13 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult

CONTACTS AND LOCATIONS:
Locations (24):
- United States (24):
  - East Bay AIDS Ctr, Berkeley, California
  - Dr Milton Estes, Mill Valley, California
  - Infectious Disease Med Group / Adult Immunology Clinic, Oakland, California
  - UCI Med Ctr, Orange, California
  - Kaiser Permanente Med Ctr, San Francisco, California
  - Santa Clara Valley Med Ctr, San Jose, California
  - Pfizer Central Research, Groton, Connecticut
  - Georgetown Univ Med Ctr, Washington D.C., District of Columbia
  - Whitman - Walker Clinic, Washington D.C., District of Columbia
  - Med Service, Miami, Florida
  - Dr Robert Wallace, St. Petersburg, Florida
  - Bay Area AIDS Consortium, Tampa, Florida
  - West Paces Clinical Research Inc, Atlanta, Georgia
  - Northwestern Univ Med School, Chicago, Illinois
  - Dr Neel French / Louis A Weiss Memorial Hosp, Chicago, Illinois
  - Oschner Clinic, New Orleans, Louisiana
  - Trinity Lutheran Hosp / Infectious Disease Clinic, Kansas City, Missouri
  - Duke Univ Med Ctr, Durham, North Carolina
  - Austin Infectious Disease Consultants, Austin, Texas
  - Central Texas Med Foundation, Austin, Texas
  - Univ of Texas Southwestern Med Ctr of Dallas, Dallas, Texas
  - Thomas Street Clinic / Baylor College of Medicine, Houston, Texas
  - Dr Gary Brewton, Houston, Texas
  - Hampton Roads Med Specialists, Hampton, Virginia

REFERENCES:
- [Background] Dunne M, Fessel J, Kumar P, Dickenson G, Keiser P, Boulos M, Mogyros M, White AC Jr, Cahn P, O'Connor M, Lewi D, Green S, Tilles J, Hicks C, Bissett J, Schneider MM, Benner R. A randomized, double-blind trial comparing azithromycin and clarithromycin in the treatment of disseminated Mycobacterium avium infection in patients with human immunodeficiency virus. Clin Infect Dis. 2000 Nov;31(5):1245-52. doi: 10.1086/317468. Epub 2000 Nov 6. PMID 11073759